CLINICAL TRIAL: NCT06353386
Title: MK-5684-01A Substudy: A Phase 1/2 Umbrella Substudy of MK-5684-U01 Master Protocol to Evaluate the Safety and Efficacy of MK-5684-based Treatment Combinations or MK-5684 Alone in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Substudy 01A: Safety and Efficacy of Opevesostat (MK-5684)-Based Treatment Combinations or Opevesostat Alone in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-5684-01A)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5684-01A; MK-5684-01A (Other: MSD); 2023-506288-33-00 (Registry Identifier: EU CT); U1111-1292-6912 (Registry Identifier: UTN); jRCT2031240224 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — olaparib; Docetaxel; cabazitaxel; fludrocortisone acetate; Dexamethasone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A1: Opevesostat (Experimental): Participants receive 5 mg of opevesostat twice daily (BID) via oral tablet plus dexamethasone 1.5 mg by oral tablets once daily (QD) and 0.1 mg fludrocortisone acetate by oral tablet QD until progression or discontinuation.
  Interventions: Drug: Opevesostat; Drug: Fludrocortisone acetate; Drug: Dexamethasone
- Arm A2: Olaparib + Opevesostat (Experimental): Participants receive 5 mg of opevesostat BID via oral tablet plus dexamethasone 1.5 mg by oral tablets QD and 0.1 mg fludrocortisone acetate by oral tablet QD, PLUS 300 mg of olaparib BID via oral tablet until progressive disease or discontinuation.
  Interventions: Drug: Opevesostat; Drug: Olaparib; Drug: Fludrocortisone acetate; Drug: Dexamethasone
- Arm A3: Docetaxel + Opevesostat (Experimental): Participants receive 5 mg of opevesostat BID via oral tablet plus dexamethasone 1.5 mg by oral tablets QD and 0.1 mg fludrocortisone acetate by oral tablet QD, PLUS 75 mg/m^2 of docetaxel once every 3 weeks (Q3W) via IV infusion, plus prednisone per approved product label BID by oral tablets until progressive disease or discontinuation.
  Interventions: Drug: Opevesostat; Drug: Docetaxel; Drug: Fludrocortisone acetate; Drug: Dexamethasone; Drug: Prednisone
- Arm A4: Cabazitaxel + Opevesostat (Experimental): Participants receive 5 mg of opevesostat BID via oral tablet plus dexamethasone 1.5 mg by oral tablets QD and 0.1 mg fludrocortisone acetate by oral tablet QD, PLUS 20 mg/m^2 of cabazitaxel Q3W via IV infusion, plus prednisone per approved product label BID by oral tablets until progressive disease or discontinuation.
  Interventions: Drug: Opevesostat; Drug: Cabazitaxel; Drug: Fludrocortisone acetate; Drug: Dexamethasone; Drug: Prednisone

INTERVENTIONS:
Drug: Opevesostat — Oral Tablet
  Other Names: MK-5684
Drug: Olaparib — Oral Tablet
  Other Names: LYNPARZA®
  Arms: Arm A2: Olaparib + Opevesostat
Drug: Docetaxel — IV Infusion
  Other Names: TAXOTERE®
  Arms: Arm A3: Docetaxel + Opevesostat
Drug: Cabazitaxel — IV Infusion
  Other Names: JEVTANA®
  Arms: Arm A4: Cabazitaxel + Opevesostat
Drug: Fludrocortisone acetate — Oral Tablet
Drug: Dexamethasone — Oral Tablet
Drug: Prednisone — Oral Tablet
  Arms: Arm A3: Docetaxel + Opevesostat; Arm A4: Cabazitaxel + Opevesostat

SUMMARY:
Substudy 01A is part of a larger research study that is testing experimental treatments for metastatic castration-resistant prostate cancer (mCRPC). The larger study is the umbrella study (U01).

The goal of substudy 01A is to evaluate the safety and efficacy of opevesostat-based treatment combinations, or as a single agent, in participants with mCRPC.

This substudy will have two phases: a safety lead-in phase and an efficacy phase. The safety lead-in phase will be used to evaluate the safety and tolerability, and to establish a recommended Phase 2 dose (RP2D) for the opevesostat-based treatment combinations. There will be no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate without small cell histology.
* Prostate cancer progression and received androgen deprivation therapy (ADT) or post bilateral orchiectomy within 6 months before screening.
* Evidence of disease progression from either, >4 weeks from last flutamide treatment, or >6 weeks from last bicalutamide or nilutamide treatment, if receiving first generation anti-androgen therapy as last treatment therapy.
* Current evidence of metastatic disease.
* Prior treatment with 1 to 2 novel hormonal agent(s) (NHA) for non-metastatic, or metastatic, hormone-sensitive prostate cancer or castration-resistant prostate cancer and have disease progression during or after treatment.
* Treatment with bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses for >4 weeks before randomization.
* Participants who experienced adverse events (AEs) due to previous anticancer therapies must have recovered to <Grade 1 or baseline.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy.
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load.
* Participants with a history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of pituitary dysfunction.
* Poorly controlled diabetes mellitus.
* Active or unstable cardio/cerebro-vascular disease, including thromboembolic events and history of stroke or transient ischemic attack within 6 months before the first dose of study intervention, history of myocardial infarction within 6 months before the first dose of study intervention, New York Heart Association Class III or IV cardiac disease or congestive heart failure, coronary heart disease that is symptomatic, or unstable angina
* History or family history of long corrected QT interval (QTc) syndrome.
* Myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or features suggestive of MDS/AML.
* History or current condition of adrenal insufficiency.
* History of (noninfectious) pneumonitis requiring steroids, or current pneumonitis.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Undergone major surgery, including local prostate intervention (except prostate biopsy) within 28 days before randomization, and has not recovered from the toxicities and/or complications.
* Is on an unstable dose of thyroid hormone therapy within 6 months prior to first dose of study intervention.
* Received a whole blood transfusion in the last 120 days before randomization (packed red blood cells and platelet transfusions are acceptable if not given within 28 days before randomization).
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities, requiring corticosteroids.
* Received a live or live-attenuated vaccine within 30 days before the first does of study intervention. Administration of killed vaccines is allowed.
* Diagnosis of immunodeficiency, or is receiving chronic systemic steroid therapy, or any other form of immunosuppressive therapy, within 7 days prior to the first dose of study intervention.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* Active infection requiring systemic therapy.
* Concurrent active HBV or HCV infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more dose-limiting toxicities (DLTs) | Up to approximately 28 days
  The following events, if considered drug related by the investigator, will be considered a DLT: Grade 4 nonhematologic toxicity (not laboratory value); Grade 4 hematologic toxicity lasting >7 days, except thrombocytopenia (Grade 4 thrombocytopenia of any duration, Grade 3 thrombocytopenia associated with clinically significant bleeding); Any nonhematologic adverse event (AE) >Grade 3 in severity should be considered a DLT (with exceptions); Any Grade 3 or Grade 4 nonhematologic laboratory value (if certain criteria are met); Febrile neutropenia Grade 3 or Grade 4; Prolonged delay (>2 weeks) in initiating treatment after the first 28 days due to study intervention-related toxicity; Missing >25% of study intervention doses as a result of drug-related AE(s) during the first 28 days; Grade 5 toxicity.
Number of participants who experience one or more adverse events (AEs) | Up to approximately 46 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to approximately 46 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Prostate-specific antigen (PSA) response rate | Up to approximately 46 months
  The Prostate-specific Antigen (PSA) response rate is the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by ≥50%. The reduction in PSA level will be confirmed by an additional PSA evaluation performed ≥3 weeks from the original response per Prostate Cancer Working Group (PCWG) criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 46 months
  The ORR is defined as the percentage of participants with complete response (CR: disappearance of all target lesions per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1); and no evidence of disease (NED) on base scan per Prostate Cancer Working Group (PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG). ORR will be assessed by Blinded Independent Central Review (BICR).
Radiographic progression-free survival (rPFS) | Up to approximately 46 months
  rPFS is defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Progression as per modified RECIST 1.1 is ≥20% increase in the sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria is the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and are persistent for ≥6 weeks. rPFS will be assessed by BICR.
Overall survival (OS) | Up to approximately 46 months
  OS is defined as the time from randomization to death due to any cause.
Duration of response (DOR) | Up to approximately 46 months
  DOR is defined as the time from first documented evidence of complete response (CR) or partial response (PR) per PCWG and RECIST 1.1 criteria until progressive disease (PD) or death. PD per RECIST 1.1 is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of a least 5 mm. PD per PCWG is the appearance of >2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and are persistent for >6 weeks. DOR will be assessed by BICR.
Time to first subsequent anticancer therapy (TFST) | Up to approximately 46 months
  TFST is defined as the time from randomization to initiation of the first subsequent anticancer therapy or death, whichever occurs first.
Time to pain progression (TTPP) | Up to approximately 46 months
  TTPP is defined as the time from randomization to pain progression based on the Brief Pain Inventory-Short Form (BPI-SF) Item 3 "worst pain in 24 hours" and by opiate analgesic use.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (77):
- United States (7):
  - UCSD Moores Cancer Center ( Site 0039), La Jolla, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0044), Los Angeles, California
  - University of Miami Hospital and Clinics, Sylvester Cancer Center-Cancer Research Services ( Site 0051), Miami, Florida
  - University of Maryland-Greenebaum Comprehensive Cancer Center ( Site 0049), Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey ( Site 0033), New Brunswick, New Jersey
  - University Hospitals Cleveland Medical Center ( Site 0043), Cleveland, Ohio
  - MEDICAL COLLEGE OF WISCONSIN-Cancer Center Clinical Trials Office ( Site 0020), Milwaukee, Wisconsin
- Australia (3):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0108), Macquarie University, New South Wales
  - Gallipoli Medical Research Ltd-GMRF CTU ( Site 0107), Greenslopes, Queensland
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0110), Melbourne, Victoria
- Canada (3):
  - Centre Hospitalier de l'Université de Montréal ( Site 0200), Montreal, Quebec
  - Jewish General Hospital ( Site 0206), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0207), Québec, Quebec
- Chile (5):
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0304), Talca, Maule Region
  - FALP ( Site 0301), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0303), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0300), Santiago, Region M. de Santiago
  - CIDO SpA-Oncology ( Site 0302), Temuco, Región del Biobío
- Colombia (5):
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0406), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 0402), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0400), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0404), Montería, Departamento de Córdoba
  - Fundación Valle del Lili-Oncology CIC ( Site 0403), Cali, Valle del Cauca Department
- Denmark (2):
  - Herlev and Gentofte Hospital ( Site 0501), Copenhagen, Capital Region
  - Aalborg Universitetshospital, Syd ( Site 0503), Aalborg, North Denmark
- Finland (3):
  - Vaasan Keskussairaala ( Site 0603), Vaasa, Pohjanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 0604), Helsinki, Uusimaa
  - Docrates Syöpäsairaala ( Site 0602), Helsinki, Uusimaa
- France (4):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0700), Strasbourg, Alsace
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 0703), Bordeaux, Aquitaine
  - Hôpital Européen Georges Pompidou-Service d'Oncologie Médicale ( Site 0702), Paris
  - Gustave Roussy ( Site 0701), Villejuif, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Heidelberg ( Site 0805), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen-Urologie ( Site 0801), Tübingen, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Site 0802), Munich, Bavaria
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0800), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf-Onkologisches Zentrum ( Site 0804), Hamburg
- Ireland (3):
  - St. Vincent's University Hospital ( Site 0901), Dublin, Dublin
  - Cork University Hospital ( Site 0902), Cork
  - Tallaght University Hospital ( Site 0900), Dublin
- Israel (3):
  - Rambam Health Care Campus-Oncology Division ( Site 1002), Haifa
  - Rabin Medical Center ( Site 1001), Petah Tikva
  - Sheba Medical Center ( Site 1000), Ramat Gan
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1102), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1103), Milan, Lombardy
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1101), Rozzano, Milano
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedal-Centro Ricerche Cliniche di Verona ( Site 1100), Verona
- Japan (4):
  - Toho University Sakura Medical Center ( Site 1201), Sakura, Chiba
  - Yokohama City University Medical Center ( Site 1203), Yokohama, Kanagawa
  - The Jikei University Hospital ( Site 1202), Mitato, Tokyo
  - Kyushu University Hospital ( Site 1204), Fukuoka
- Auckland City Hospital ( Site 1333), Auckland, New Zealand
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1402), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 1400), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 1405), Gdansk, Pomeranian Voivodeship
- South Korea (3):
  - Asan Medical Center-Oncology ( Site 1500), Songpagu, Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1502), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1501), Seoul
- Spain (5):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 1603), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1600), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1602), Barcelona
  - Hospital General Universitario Gregorio Marañón ( Site 1601), Madrid
  - Hospital Clinico San Carlos-Oncology Department ( Site 1604), Madrid
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 1704), Kaohsiung Niao Sung Dist, Kaohsiung
  - China Medical University Hospital ( Site 1703), Taichung
  - Taipei Veterans General Hospital ( Site 1701), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Medical Oncology ( Site 1702), Taoyuan District
- Turkey (Türkiye) (5):
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 1802), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1800), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 1801), Ankara
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1804), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1803), Istanbul
- United Kingdom (5):
  - Addenbrooke's Hospital ( Site 1902), Cambridge, Cambridgeshire
  - The Beatson West of Scotland Cancer Centre ( Site 1904), Glasgow, Glasgow City
  - Royal Preston Hospital-Lancashire Clinical Research Facility ( Site 1900), Preston, Lancashire
  - University College London Hospital ( Site 1905), London, London, City of
  - Queen Elizabeth Hospital Birmingham ( Site 1903), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26115&tenant=MT_MSD_9011